CLINICAL TRIAL: NCT03161743
Title: Calculation of Platelet-rich Plasma Preparation Yield From Baseline CBC Platelet Count
Brief Title: Calculation of Platelet-rich Plasma Preparation Yield
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Harrison, Theodore, M.D. (Individual)
Responsible Party: Principal Investigator, Theodore Harrison, MD, Principal Investigator, Harrison, Theodore, M.D.
Other Study IDs: PRP Platelet Yield
Record Dates: First submitted 2017-05-18; First posted 2017-05-22 (Actual); Last update posted 2017-08-10 (Actual); Status verified 2017-08

CONDITIONS: Platelet-rich Plasma Production
Keywords: platelet-rich plasma; platelet
MeSH Terms: interventions — Phlebotomy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: venipuncture — blood draw for the purpose of determining the platelet concentration in PRP

SUMMARY:
This is a study to determine 1) the consistency of platelet-rich plasma produced by several methods, and 2) whether the platelet content of platelet-rich plasma can be accurately estimated from a baseline CBC platelet count.

DETAILED DESCRIPTION:
In the first phase of this study a baseline CBC platelet count will be performed on each subject and then platelet-rich plasma (PRP) prepared from the same blood sample by six different methods. The platelet count will be measured in each PRP preparation and compared to the CBC platelet count to determine the platelet yield for each method.

In the second phase of the study a baseline CBC platelet count will be performed on each subject and then platelet-rich plasma (PRP) prepared from the same blood sample by six different methods. The CBC platelet count will be used to calculate the estimated platelet content of each sample/method based on the platelet yields determined in the first phase. The platelet count will be measured in each PRP preparation and compared to the estimated platelet content to determine the predictive accuracy for each method.

ELIGIBILITY:
Inclusion Criteria:

* English speaking

Exclusion Criteria:

* platelet count < 150,000
* platelet count > 350,000
* History of blood disorder
* History of altered platelet function
* History of chemotherapy or radiation therapy

Ages: 21 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: normal adults
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2017-06-30 (Actual); Primary Completion 2018-05-31 (Estimated); Study Completion 2018-05-31 (Estimated)

PRIMARY OUTCOMES:
Platelet yield | within 8 hours of blood draw
  the number of platelets in a PRP sample as a percentage of the number of platelets in the blood from which the PRP was prepared.
Platelet yield estimate accuracy | within one month of final data collection
  standard deviation of the difference between the estimated platelet yield and the actual platelet yield.

CONTACTS AND LOCATIONS:
Overall Officials: Theodore E Harrison, Principal Investigator — Theodore Harrison
Locations (1):
- Theodore E Harrison, Sidney, British Columbia, Canada

IPD SHARING:
Plan to Share IPD: No